CLINICAL TRIAL: NCT03046771
Title: Randomized Controlled Trial Evaluating Efficacy of EMS Providers Performing Discharge Comprehension and Home Fall Hazard Assessments
Brief Title: Transport PLUS Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 14-1842; 1R03AG050917-01 (NIH)
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Fall, Accidental; Fall; Hospital Readmission; Emergency Medical Services
Keywords: falls; readmissions; emergency department visits; transitions of care
MeSH Terms: interventions — Parturition; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transport PLUS group (Experimental): EMTs randomized to the Transport Plus group will view a 60-minute training video and then complete a 60-minute simulation training exercise on how to conduct the home fall hazard assessment (FHA) and the discharge comprehension assessment (DCA) and how to complete the FHA and DCA checklists. The FHA involves performing a visual assessment of the home environment and noting certain fall hazards. The DCA involves engaging the patient or caregiver in a conversation to assess their level of understanding of the elements of the discharge instructions. The Transport Plus EMTs will offer to perform the FHA and DCA for all transports of patients aged 65 or older, who are being transported from The Mount Sinai Hospital to a private residence
  Interventions: Behavioral: Transport PLUS group
- Routine Care (No Intervention): Providers randomized to routine care will not be trained on the FHA or DCA or the completion of the checklists. All EMTs in both groups (Transport Plus and standard education), will be asked to answer some demographic questions and will be trained to collect responses to 3questions commonly used to assess a patient's risk of falling and to collect best contact information for phone follow up from patients or their caregivers and to obtain permission for a follow-up phone call from research personnel.

INTERVENTIONS:
Behavioral: Transport PLUS group — The Transport Plus EMTs will offer to perform the FHA and DCA for all transports of patients aged 65 or older, who are being transported from The Mount Sinai Hospital to a private residence.
  Arms: Transport PLUS group

SUMMARY:
Hypothesis: 'Transport PLUS,' a low cost, easily generalizable intervention performed by Emergency Medical Technicians while transporting a patient home from the hospital, can improve transitions of care and improve patient safety following hospitalization as measured by decreased rates of falls and reduced rates of return to the hospital.

DETAILED DESCRIPTION:
The moment of transition between the hospital and the home is susceptible to lapses in quality and loss of key information regarding a patient's care. An increasing amount of attention is being given to improving the transition of care by targeting factors that contribute to return Emergency Department (ED) visits and readmissions. Following a hospitalization, as many as 40% of patients over age 60 will experience a fall in the subsequent six months and 76% of older adult patients are uncertain about their follow-up care plan. Patients transported home by ambulance following an ED visit were found to have a significantly higher rate of return ED visits at 30 days then overall rates for older adult ED patients (27.8% vs. 11.5%).

In response to these challenges, the researcher's study group developed and piloted an innovative care model known as "Transport PLUS" in which specially trained emergency medical technicians (EMTs) who are already transporting an older adult (65+ years in age) patient home from the ED add to their service two simple interventions - a home fall hazard assessment (FHA) and a discharge comprehension assessment (DCA). Both interventions are facilitated and measured using a checklist developed through a systematic review of the literature and existing tools, and later refined through EMT and patient focus groups.

This study will test the hypothesis that 'Transport PLUS,' a low cost, easily generalizable intervention, can improve transitions of care and improve patient safety following hospitalization as measured by decreased rates of falls and reduced rates of return to the hospital.

The researchers will conduct a pilot cluster randomized controlled trial comparing the Transport PLUS intervention to standard care in a population of older adult patients being discharged from the hospital. The researchers will randomize EMS providers to either perform Transport PLUS (the intervention) or to provide routine transport. It is estimated that approximately 400 patients over age 65 will be transported home from the study hospital by participating providers during the study enrollment period. Patient participants will receive Transport PLUS (n=200) or routine care (n=200) as determined by the transporting provider. Primary outcomes will be the rate of falls in the 3 months following hospitalization and 3-day and 30-day return ED visits (with or without a hospitalization). Process measures will include removal of fall hazards at 3 months and compliance with discharge instructions. Extending beyond the grant period, the researchers intend to follow the cohort for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

Emergency Medical Technicians (EMTs) are eligible to participate in study if

* employed by Hunter EMS
* over the age of 18 years, and
* certified as an EMT in New York State.

Patient participants are eligible if

* over the age of 65 years
* being discharged from the study hospital, and
* being transported directly to home.

Exclusion Criteria:

* EMTs who expect to leave the job in less than 1 year
* EMTs who have been previously trained in Transport PLUS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Rate of falls | up to 3 months
  Rate of falls following transport home by ambulance
Rate of return ED visits | 30 days
  Rate of return ED visits following transport home by ambulance

SECONDARY OUTCOMES:
Rate of falls | up to 12 months
Rate of return ED visits | 3 days
  Numbers of patients with ED visits within 3 days of participation in study intervention or control arm.
Readmission | up to 90 days
  Numbers of patients with readmissions after study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Munjal, MD,MPH,MSCR, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No